CLINICAL TRIAL: NCT03711097
Title: The Effectiveness of Resin-Modified Glass Ionomer Varnish in Preventing White Spot Lesions During Fixed Appliance Orthodontic Therapy
Brief Title: Effectiveness of Resin-Modified Glass Ionomer Varnish in Preventing White Spot Lesions in Fixed Appliance Orthodontia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study not initiated
Sponsor: University of Nebraska (Other)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0548-18-FB
Record Dates: First submitted 2018-10-14; First posted 2018-10-18 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: White Spot Lesion

STUDY DESIGN:
Intervention Model Description: Split mouth study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (No Intervention): Upper left or right central and lateral incisor
- Varnish Intervention (Experimental): Upper central and lateral incisor contralateral to control upper central and lateral incisor
  Interventions: Drug: Vanish XT Dental Varnish

INTERVENTIONS:
Drug: Vanish XT Dental Varnish — Varnish will be applied to the front surface of the intervention upper central and lateral incisors
  Other Names: resin-modified glass ionomer
  Arms: Varnish Intervention

SUMMARY:
This is a prospective study to determine the effects of resin-modified glass ionomer (RMGI) on the prevention of white spot lesion (WSL) development during fixed appliance orthodontic treatment. WSLs are the beginning stages of cavity formation on teeth and RMGI is a preventative material placed on teeth. The RMGI will be applied at the initial bonding appointment when braces are put on. RMGI will be applied to some participant's teeth while others will not receive the varnish treatment. Patients will be given standardized oral hygiene instructions. At six months, the RMGI will be reapplied to the same teeth that received the original RMGI application. The development of WSLs will be assessed both by photographs and visual assessment as well as utilizing laser technology to assess the level of enamel demineralization via a dental scanner called the Canary System. Participants will be examined at 3-month intervals for a total of nine months to one year to determine if application of RMGI during fixed appliance orthodontic therapy is effective in preventing the development of WSLs.

DETAILED DESCRIPTION:
This study is a prospective study to assess the effects of resin-modified glass ionomer (RMGI) on the prevention of white spot lesion (WSL) development during fixed appliance orthodontic treatment. WSLs are the beginning stages of cavity formation on teeth and RMGI is a material that is placed on the teeth to prevent WSLs. Patients will be recruited from the UNMC College of Dentistry Orthodontic Clinic who have been treatment planned to undergo fixed appliance therapy to include the maxillary central and lateral and central incisor teeth, which are the upper front four teeth in the mouth. In order to be included in this study, these teeth need to be fully erupted and planned to have braces on their front surfaces for a minimum of six months. The RMGI will be applied at the initial bonding appointment, which is the appointment that the subject receives their braces, to the labial surfaces of the teeth either to the right or left side central and lateral incisor. The control teeth will be the upper central and lateral incisors that do not receive the varnish treatment. Assignment of the left or right side will be randomized to obtain equal numbers of left and right-sided RMGI applications, mitigating the potential effects related to the handedness of the patients. The patients will be given standardized oral hygiene instructions and will be seen in follow up at 3-month intervals. At the 6-month mark, the RMGI will be reapplied to the same teeth that received the original RMGI application. At the initial bonding appointment and at each 3-month interval following, the development of WSLs will be assessed both by photographs and visual assessment as well as utilizing laser technology to assess the level of enamel demineralization via a dental scanner called the Canary System. Measurements and application of the RMGI will be performed by an individual examiner and a random subset of measurements will be re-measured after adequate washout time to ensure high intra-examiner reliability. Photographs will be assessed by examiners that have been blinded to the teeth receiving treatment. The goal of this study is to have the patients examined at 3-month intervals for a total treatment time of nine months to one year to ascertain if application of RMGI to the labial surfaces of the central and lateral incisor teeth during fixed appliance orthodontic therapy is effective in preventing the development of WSLs.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in research project
* Age ≥ 10 years old, fully erupted maxillary central and lateral incisors
* treatment time with fixed appliances estimated to be at least 6 months

Exclusion Criteria:

* Presence of peg lateral maxillary incisors
* Presence of one or more significant WSLs on maxillary incisors prior to orthodontic therapy
* Restorations covering a significant portion of the labial surfaces of the maxillary incisors
* Unerupted maxillary incisors, presence of uncontrolled caries
* Craniofacial Syndromic patients and patients with cleft lip and/or palate
* Pregnant or breast-feeding patients

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Development of White Spot Lesion on the Labial Surface of the Upper Central and/or Lateral Incisors | 6-9 months
  The development of white spot lesion in subjects will be determined by photographs that are evaluated for white spot lesions by experienced orthodontists as well as by objectively measuring the level of demineralization of the teeth based on dental scanning technology (The Canary System). The Canary System gives a numerical score based on the level of demineralization of the tooth and indicates if demineralization is progressing or improving over time.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Herman, DDS, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No